CLINICAL TRIAL: NCT00530049
Title: Measuring Patient Satisfaction With Facial Appearance: Development and Validation of a New Patient-Reported Outcome Measure
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); McMaster University (Other); The New School for Social Research (Other); University College, London (Other); Yeshiva University (Other)
Responsible Party: Sponsor
Other Study IDs: 07-098; MSKCC-07098
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Head and Neck Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; metastatic squamous neck cancer with occult primary; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; salivary gland cancer; tongue cancer; 07-098
MeSH Terms: conditions — Head and Neck Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- questionnaires: The purpose of this study is to develop a PRO instrument that measures quality of life as relates to facial appearance after head and neck cancer reconstruction surgery and after dermatologic surgery for patients with cutaneous skin cancers. . To develop this measure, we will adhere to the following sequential steps recommended by quality of life experts. Thus, the study will have three parts:
  * Questionnaire content generation and development of preliminary instrument
  * Field-testing the preliminary questionnaire with item reduction and development of final questionnaire
  * Psychometric evaluation of final questionnaire
  Interventions: Other: questionnaire administration; Procedure: assessment of therapy complications; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment

INTERVENTIONS:
Other: questionnaire administration
Procedure: assessment of therapy complications
Procedure: psychosocial assessment and care
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Developing a questionnaire that patients can use to assess their quality of life related to the appearance of their face after surgery may help doctors plan the best treatment for patients undergoing surgery and reconstruction for head and neck cancer in the future.

PURPOSE: This clinical trial is developing a questionnaire for assessing quality of life related to facial appearance in patients who have undergone or are planning to undergo surgery and reconstruction for head and neck cancer; and after dermatologic surgery for patients with cutaneous skin cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop and validate a new patient-reported outcome measure of quality of life related to facial appearance following oncologic head and neck resection and reconstruction.

OUTLINE:

* Part 1 (questionnaire content generation and development of preliminary instrument [post-operative patients only]): Patients undergo semi-structured interview with a trained interviewer and answer open-ended questions. Statements concerning facial appearance post-resection and reconstruction are extracted to generate items for the preliminary instrument. The preliminary instrument is developed from review of the literature, qualitative interviews with patients, and expert opinion (head and neck surgeons, reconstructive surgeons, and other relevant health care providers, including nurse clinicians). The instrument is then pre-tested on a small sample of patients via mail to clarify ambiguities in the wording of items, confirm appropriateness, and determine acceptability and completion time.
* Part 2 (field-testing with item reduction and development of final rating scale): Post-operative patients complete 2 copies of the preliminary questionnaires in the mail or clinic approximately 2 weeks apart. Pre-operative patients complete the questionnaire prior to surgery (during preoperative appointment) and again at least 1 month after surgery (via mail). Data are analyzed to determine the most valid grouping of items into measurement scales for development of the final instrument.
* Part 3 (psychometric evaluation of the patient-reported outcome questionnaire): Post-operative patients complete 2 copies of the questionnaires in clinic or by mail approximately 2 weeks apart. They also complete several other well-established, validated instruments used to measure patient-reported quality of life and symptomatology in order to aid in the evaluation of convergent and discriminant validity. Pre-operative patients complete the final questionnaire prior to surgery (during preoperative appointment) and again at least 1 month after surgery by mail or in clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 99 years.
* Patients who have altered facial appearance secondary to an oncologic head and neck surgical resection and reconstruction. Reconstruction will be defined as complex linear closures, skin grafts, local flaps or free tissue transfer (oncologic Post-op cohort).
* Patients who have undergone cosmetic plastic surgery procedures to the head and neck unrelated to a diagnosis of cancer (non-oncologic Post-op cohort).
* Patients with cutaneous skin cancers of the head and neck region treated in the dermatologic surgery setting (dermatology Post-op cohort)
* Patients who have completed surgery at MSKCC between 1 week to 7 years ago (Post-op cohorts).
* Patients who have completed facial surgery 6 weeks (+/- 1 week) ago (early postoperative subset-Phase I).
* Patients who are scheduled to undergo oncologic head and neck resection and reconstruction with anticipated altered facial appearance (Pre-op).
* Patients who are scheduled to undergo dermatologic surgery due to diagnosis cutaneous skin cancers of the head and neck region (dermatology Pre-op cohort)

Exclusion Criteria:

* Active psychiatric illness, cognitive or sensory impairment that in the opinion of the investigator is severe enough to preclude participation in the study.
* Moderate to severe cognitive impairment.
* Blindness.
* Physical impairment that may prevent the respondent from filling out the paper and pencil survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC), or specified plastic surgeon at outside institution.
Sampling Method: Non-Probability Sample
Enrollment: 1745 (Estimated)
Dates: Start 2007-08-14 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
Development of patient-reported outcome measure of quality of life related to facial appearance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L. Pusic, MD, MHS, Principal Investigator — Memorial Sloan Kettering Cancer Center; Peter G. Cordeiro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (2):
  - New School for Social Research, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario, Canada
- University College of London Hospitals, London, England, United Kingdom

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm